CLINICAL TRIAL: NCT06279949
Title: Implementation of Confidential Care to Increase Adolescent HIV Testing in Pediatric Primary Care Settings
Brief Title: Confidential Care and Adolescent HIV Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 2000036999; K01MH136929 (NIH)
Record Dates: First submitted 2024-02-19; First posted 2024-02-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hiv
Keywords: Confidential care; Pediatrics; HIV testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- No provider training or clinic protocols (No Intervention): This clinic will not receive training on state-specific laws regulating minors' access to confidential HIV testing or implementation of new protocols to support confidential care provision.
- Clinic protocols (Active Comparator): This clinic will receive training on navigating new protocols to support confidential care provision.
  Interventions: Behavioral: Clinic protocols
- Provider training (Active Comparator): This clinic will receive training on state-specific laws regulating minors' access to confidential HIV testing.
  Interventions: Behavioral: Provider training
- Provider training and clinic protocols (Active Comparator): This clinic will receive training on state-specific laws regulating minors' access to confidential HIV testing and navigating new protocols to support confidential care provision.
  Interventions: Behavioral: Provider training; Behavioral: Clinic protocols

INTERVENTIONS:
Behavioral: Provider training — Clinics randomized to a condition involving provider training will receive training on state-specific laws regulating minors' access to confidential HIV testing.
  Arms: Provider training; Provider training and clinic protocols
Behavioral: Clinic protocols — Clinics randomized to a condition involving the implementation of new clinic protocols to support confidential care provision will receive training on navigating the new protocols.
  Arms: Clinic protocols; Provider training and clinic protocols

SUMMARY:
The purpose of this study is to assess the feasibility and acceptability of structural intervention components to increase adolescent HIV testing uptake by improving the implementation of confidential care as standard practice in pediatric primary care.

DETAILED DESCRIPTION:
This pilot study will evaluate a multicomponent structural intervention to increase adolescent HIV testing uptake by improving the implementation of confidential care as standard practice in pediatric primary care settings. The objectives of the study are to: (a) evaluate feasibility, acceptability, and other implementation outcomes (e.g., reach); (b) assess change in HIV testing uptake; and (c) determine the combination of structural intervention components to be further evaluated in a future full-scale optimization trial. These objectives will be achieved through a pilot optimization trial; the trial will follow a full factorial experimental design with data collection at three time points over a 12-month period.

During the 6-month pre-intervention period, baseline measures will be assessed extracting electronic health record (EHR) data on the number of adolescent patients who were screened for, accepted, and received results of HIV testing. During the 6-month intervention period, clinics will be randomized to one of four experimental conditions based on the following two factors: (1) provider training; (2) implementation of clinic protocols to support confidential care provision. Clinics randomized to a condition involving provider training will receive training on state-specific laws regulating minors' access to confidential HIV testing. Clinics randomized to a condition involving the implementation of clinic protocols will receive training on navigating the new protocols. Measurement of intervention and implementation processes and outcomes will be guided by the five dimensions of the RE-AIM Framework: reach, efficacy, adoption, implementation, and maintenance. During the 6-month post-intervention period, EHR data will be used to assess the change in HIV testing uptake over the study period.

ELIGIBILITY:
The intervention occurs at the clinic-level and so the enrolled participant is a pediatric primary care clinic. The patient-level outcome (i.e., change in HIV testing uptake) will be collected based on the following eligibility criteria:

Inclusion Criteria:

- 13-17 years old

Exclusion Criteria:

* <13 years old
* >17 years old

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility, defined as the extent to which structural intervention components to improve confidential care implementation can be successfully carried out in pediatric primary care settings | 6 months
  Feasibility will be measured with the Feasibility of Intervention Measure, a self-reported four-item measure with established reliability and validity. Item responses range from 1="completely disagree" to 5="completely agree." Scores are created by averaging responses. Score values range from 1 to 5, with higher scores indicating greater feasibility.
Acceptability, defined as the perception among pediatric primary care clinic leadership and providers that structural intervention components to improve confidential care implementation are agreeable or satisfactory | 6 months
  Acceptability will be measured with the Acceptability of Intervention Measure, a self-reported four-item measure with established reliability and validity. Item responses range from 1="completely disagree" to 5="completely agree." Scores are created by averaging responses. Score values range from 1 to 5, with higher scores indicating greater acceptability.
Change in HIV testing uptake | Baseline, 12 months
  Change in HIV testing uptake will be assessed as the difference in the number of adolescent patients who were screened for, accepted, and received results of HIV testing during the 6-month pre-intervention period compared to the 6-month post-intervention period.

SECONDARY OUTCOMES:
Reach, defined as the number of adolescent patients who receive confidential care | 6 months
  Reach will be assessed through a brief online survey to be self-administered by providers after each visit with an adolescent patient.
Adoption, defined as the proportion of pediatric primary care providers who have time alone with and/or provide confidentiality assurances to adolescent patients | 6 months
  Adoption will be assessed through a brief online survey to be self-administered by providers after each visit with an adolescent patient.
Implementation, defined as pediatric primary care provider fidelity to confidential care provision | 6 months
  Implementation will be assessed through a brief online survey to be self-administered by providers after each visit with an adolescent patient.
Maintenance, defined as the extent to which confidential care is provided and adolescent patients are screened for, accept, and receive results of HIV testing 6-months post-intervention | 12 months
  Maintenance will be assessed through a brief online survey to be self-administered by providers after each visit with an adolescent patient and the number of adolescent patients who were screened for, accepted, and received results of HIV testing during the 6-month post-intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Aivadyan, Principal Investigator — Yale University

IPD SHARING:
Plan to Share IPD: No